CLINICAL TRIAL: NCT02588781
Title: Pemetrexed Alone as Salvage Treatment in Metastatic Colorectal Cancer Patients Who Were Failed After Standard Chemotherapy: A Phase II Single Arm Prospective Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-071
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental): Pemetrexed 500 mg/m2 IV Q 3 weeks
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Alimta 500mg/m2 + NS 100ml IV infusion for 10mins Every 3weeks
  Other Names: Alimta

SUMMARY:
Pemetrexed is an anticancer agent that exerts its action by disrupting crucial folate-dependent metabolic processes essential for cell replication. In vitro studies have shown that pemetrexed behaves as a multitargeted antifolate by inhibiting thymidylate synthase (TS), dihydrofolate reductase (DHFR), and glycinamide ribonucleotide formyltransferase (GARFT), which are key folate-dependent enzymes for the de novo biosynthesis of thymidine and purine nucleotides.Pemetrexed is used as a standard therapeutic agent for lung cancer, pleural mesothelioma, peritoneal mesothelioma.In addition to these effective anti-cancer effect, Pemetrexed is not severe side effects of the medicine.

Pemetrexed has been research in colon cancer. Zhang, etc., demonstrated the anti-cancer effect of Pemetrexed in human colon cancer Cells.

Although sometimes made also two or more clinical studies, Pemetrexed was reported 15-17% of the treatment response rate in these two studies.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 20 years of age.
2. Written and voluntary informed consent understood, signed and dated.
3. They must have refractory or progressive colorectal cancer for which there is no further curative therapy available.
4. Subject able to adhere to the study visit schedule and other protocol requirements.
5. ECOG 0-2
6. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
7. Must have a life expectancy of 3 months or more
8. Demonstrate adequate organ function
9. Negative urine or serum pregnancy test within 28 days of study treatment
10. Be willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality for assessment of biomarker status.

Exclusion Criteria:

1. ECOG ≥ 3
2. History of malignancy in the last 5 years.
3. Subject has known historical or active infection with HIV, hepatitis B, or hepatitis C.
4. Breast-feeding or pregnant female
5. Patients can not the administration of Folic acid or Vitamin B12.
6. Before treatment with Pemetrexed.
7. Patients who can not swallow oral medication.
8. The most recent treatment with the clinical trial for the drug for 14 days prior to enrollment.
9. Systemic chemotherapy within three weeks after the administration of the last before the test treatment, radiation therapy patients who had been administered.
10. Except for the hair loss, it is induced before cancer treatment, all of toxicity in progress (> CTCAE1 grade).
11. Upper GI bleeding within registration before 4 weeks of Bowel obstruction or CTCAE3 or 4 grade.
12. Subject who experienced a recent myocardial infarction, including severe/unstable angina pectoris, coronary/peripheral artery bypass graft, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality, significant or uncontrolled cardiovascular disease CHF, and cerebrovascular accident or transient ischemic attack, or seizure disorder in the past year.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 2 years

SECONDARY OUTCOMES:
overall survival | 2 years
progression free survival | 2 years
Number of subjects with Adverse Events as a measure of safety and Tolerability | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea